CLINICAL TRIAL: NCT02408263
Title: Electrical Skin Conductance Monitoring as an Assessment of Post Operative Pain Scores
Status: Completed | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Oslo University Hospital (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 10106
Record Dates: First submitted 2015-02-17; First posted 2015-04-03 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Arthroplasty, Replacement, Hip; Threonine; Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Total Hip Replacement (THR) and Total Knee Replacement (TKR): 25 patients receiving a THR and 25 patients receiving aTKR. The investigators are using Skin Conductance Algesimeter (SCA) to measure pain by analyzing changes in skin conductance.
  Interventions: Procedure: Total Hip Replacement (THR) and Total Knee Replacement (TKR)

INTERVENTIONS:
Procedure: Total Hip Replacement (THR) and Total Knee Replacement (TKR) — Total Hip Replacement is a surgical procedure where the cartilage and bone of the hip joint is replaced with artificial materials. Total Knee Replacement involves replacement of all three compartments of the knee the medial, the lateral and patellofemoral compartment.

SUMMARY:
Pain has been defined as a subjective experience. Various pain assessment tools, (such as NRS) have been developed and validated to objectively monitor and treat pain. There are certain patient populations, in whom, the current pain assessment tools cannot be used effectively due to communication problems such as cognitively impaired patients. In the US, the Joint Commission on Accreditation of Healthcare Organizations (JCAHO) has made it mandatory to monitor and treat pain. In the absence of reliable pain assessment tools that would objectively measure pain, there is also risk of under treatment and overtreatment of pain that may lead to negative outcomes. Therefore, a monitor that is able to predict pain levels objectively, will help to achieve above goals. The investigators are using Skin Conductance Algesimeter (SCA) to measure pain by analyzing changes in skin conductance.

DETAILED DESCRIPTION:
Pain was defined as the fifth vital sign, and assessment and treatment of pain were introduced as a mandatory standard. This directive has improved pain management and patient satisfaction, but it has also increased the incidence of opioid-related side effects including respiratory depression with fatal outcomes. The most accepted pain assessment is the patients' self-report of their pain. Various pain assessment tools, such as the numeric rating scale (NRS), have been developed and validated. The self-report of pain is defined as the gold standard even though it may be influenced by anxiety, level of education, employment status, age and sex. The NRS is reported to be more clinically applicable than the visual analogue scale (0-100mm) specifically in elderly and in patients on opioids.The current self-report assessment tools cannot be used effectively in certain patient populations who are unable to report their pain such as cognitively impaired patients, sedated patients and children. In this group of patients, there is a risk of inadequate or overtreatment of pain which in turn may lead to negative outcomes. When patients cannot report their pain, observational and physiological parameters are used. Therefore, a monitor to objectively assess the pain would be clinically valuable. An ideal monitor would be non-invasive, fast-reacting, continuous (real-time), sensitive and specific to assess pain.

The Skin Conductance Algesimeter (SCA) measures skin sympathetic nerve activity mirrored by variations in skin conductance responses (SCR) on the palmar side of the hand. Each time the skin sympathetic nervous system is activated, the palmar and plantar sweat glands fill up with sweat. Due to electrolytes present in sweat, the skin resistance decreases and the skin conductance increases. The reabsorption of the sweat in the sweat glands reverses this process, and leads to a decrease in skin conductance. SCR can be monitored by SCA and this response is directly linked to skin sympathetic nerve activity. The number of SCR is a measure of how often the skin sympathetic nerves fire. The numbers of SCR increase during emotionally stressful stimuli like moderate-severe pain, and this is different than the painless or mild pain conditions.

To examine how the SCR is influenced by stimuli other than pain postoperatively, it is important that SCR is studied in the absence of moderate-severe pain.The goal of this study is to evaluate the correlation of SCR with emotional stressors other than pain such as: anxiety, nausea, and intellectual task performance. We hypothesized that SCR would not show a significant positive correlation with emotional stressors other than pain, thereby will increase the specificity of SCR as a viable physiological monitor for the assessment of moderate-severe pain postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral THR and TKR who are between the ages of 18 and 85 regardless of the anesthesia and postoperative analgesia type.
* Patients participating in other studies may participate in this study as well
* Patients with Motor Activity Assessment Scale (MAAS) Score of 3 and 4

Exclusion Criteria:

* Age <18, >85
* History of chronic pain as defined by use of long acting opioid medication > 6 months duration.
* MAAS Score of <3 and >4.
* Anticholinergic agent use
* Patients with the following conditions:

Autonomic neuropathy

* Pacemaker/AICD
* Burn patients or patients with severe dermatologic conditions (as defined by skin conditions causing further pain to patients that actively has to be treated)
* Allergy to adhesive tape
* Communication barriers
* Bilateral Procedures
* Patient with diagnosis of
* Dysautonomia
* Sympathetic dysfunction such as: Raynaud disease, Buerger disease
* Disorders of sweating such as: Acquired idiopathic generalized anhidrosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery for unilateral Total Hip Replacement and Total Knee Replacement.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-11; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Semih Gungor, MD, Principal Investigator — Hospital for Special Surgery, New York

REFERENCES:
- [Background] Devlin JW, Boleski G, Mlynarek M, Nerenz DR, Peterson E, Jankowski M, Horst HM, Zarowitz BJ. Motor Activity Assessment Scale: a valid and reliable sedation scale for use with mechanically ventilated patients in an adult surgical intensive care unit. Crit Care Med. 1999 Jul;27(7):1271-5. doi: 10.1097/00003246-199907000-00008. PMID 10446819
- [Background] Kunimoto M, Kirno K, Elam M, Wallin BG. Neuroeffector characteristics of sweat glands in the human hand activated by regular neural stimuli. J Physiol. 1991 Oct;442:391-411. doi: 10.1113/jphysiol.1991.sp018799. PMID 1798033
- [Background] Storm H, Shafiei M, Myre K, Raeder J. Palmar skin conductance compared to a developed stress score and to noxious and awakening stimuli on patients in anaesthesia. Acta Anaesthesiol Scand. 2005 Jul;49(6):798-803. doi: 10.1111/j.1399-6576.2005.00665.x. PMID 15954962

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Hip Replacement (THR): Patients undergoing unilateral hip replacement (THR) that are between the ages of 18 and 85. Patients with the condition of chronic pain, using long acting opioid medication >6 months will be excluded.
- Total Knee Replacement (TKR): Patients undergoing unilateral knee replacement (TKR) that are between the ages of 18 and 85. Patients with the condition of chronic pain, using long acting opioid medication >6 months will be excluded.
Period: Overall Study
Arm/Group | Total Hip Replacement (THR) | Total Knee Replacement (TKR)
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | THR and TKR
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Rating Scale
Description: Numeric Pain Rating Scale, 0 (no pain) to 10 (worst pain)
Time Frame: Baseline, Postoperative day 1, Postoperative Day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | THR and TKR
Number analyzed (Participants) | 50
units on a scale
  Baseline | 2.0 (2.2)
  Postoperative day 1 | 2.7 (2.4)
  Postoperative day 2 | 2.9 (2.0)

2. Primary Outcome: Skin Conductance Response
Description: A skin conductance response is defined as a minimum followed by a maximum in conductance values micro Siemens (mS).
Time Frame: Baseline, Postoperative day 1, Postoperative day 2
Measure: Mean (Standard Deviation); unit: micro Siemens (mS)
Groups:
- Total Hip Replacement (THR) and Total Knee Replacement (TKR): 25 patients receiving a Total Hip Replacement and 25 patients receiving a Total Knee Replacement. The investigators are using Skin Conductance Algesimeter (SCA) to measure pain by analyzing changes in skin conductance.
  THR and TKR: Total Hip Replacement is a surgical procedure whereby the diseased cartilage and bone of the hip joint is surgically replaced with artificial materials. Total Knee Replacement is a procedure which involves replacement of all three compartments of the knee (the medial compartment (inside aspect of the knee), the lateral compartment (outside of the knee) and the patellofemoral compartment (in front of the knee)).
Arm/Group | Total Hip Replacement (THR) and Total Knee Replacement (TKR)
Number analyzed (Participants) | 50
micro Siemens (mS)
  Baseline | 0.13 (0.15)
  Postoperative day 1 | 0.08 (0.12)
  Postoperative day 2 | 0.11 (0.12)

3. Secondary Outcome: Nausea
Description: Nausea was assessed by patients' self-report on their level of nausea on a 0-3 scale: 0=No nausea; 1=Mild nausea; 2=Moderate nausea; 3=Severe nausea.
Time Frame: Baseline, Postoperative day 1, Postoperative day 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Total Hip Replacement (THR) and Total Knee Replacement (TKR)
Number analyzed (Participants) | 50
units on a scale
  Baseline | 0.16 (0.51)
  Postoperative day 1 | 0.20 (0.60)
  Postoperative day 2 | 0.16 (0.51)

ADVERSE EVENTS:
Arm/Group | THR and TKR
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes